CLINICAL TRIAL: NCT04127253
Title: Evaluation of the Hypoalgesic Effects of Transcranial Direct Current (tDCS) in Combination With Motion Representation Tools in Healthy Subjects: a Double-blind Randomized Placebo-controlled Trial.
Brief Title: Evaluation of the Hypoalgesic Effects of Transcranial Direct Current (tDCS) in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: uammadrid
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Pain Modulation
Keywords: Motor imagery; Transcranial direct current stimulation; Action observation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- transcranial direct current plus Brain training tools (Experimental): 20 minutes of transcranial direct current stimulation along with the application of motor imagery and action observation
  Interventions: Device: Sooma transcranial direct current stimulation device plus Brain training tools
- Placebo transcranial direct current plus Brain training tools (Placebo Comparator): A placebo intervention of direct transcranial stimulation being active during 15 seconds and then it will be turned off the rest of the time until 20 minutes. This group will also carry out the training of action observation and motor imagery.
  Interventions: Device: Placebo Sooma transcranial direct current stimulation deviceplus Brain training tools
- Brain training tools in isolation (Sham Comparator): This group will act as a control, they will only carry out the training of action observation and motor imagery.
  Interventions: Behavioral: Brain training tools in isolation

INTERVENTIONS:
Device: Sooma transcranial direct current stimulation device plus Brain training tools — This group will carry out an observation training of actions and motor imagery in combination with the stimulation of the transcranial direct current.
  Arms: transcranial direct current plus Brain training tools
Device: Placebo Sooma transcranial direct current stimulation deviceplus Brain training tools — This group will carry out an observation training of actions and motor imagery in combination with the placebo stimulation of the transcranial direct current, where it will be acrtivo during 15 seconds and then it will be turned off during the rest of the intervention.
  Arms: Placebo transcranial direct current plus Brain training tools
Behavioral: Brain training tools in isolation — This group will act as a control, they will only carry out the training of action observation and motor imagery.
  Arms: Brain training tools in isolation

SUMMARY:
The main objective of this research is to evaluate and quantify hypoalgesic effects caused by imagination and observation with or without the presence of transcranial direct current (tDCS) in healthy participants. The secondary objective of this research is to evaluate the possible relationships between hypoalgesic effects and different physical and cognitive variables such as the ability to generate motor mental images, mental chronometry and levels of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic participants
* men and women aged 18 to 65 years

Exclusion Criteria:

* insomnia
* nausea
* headache
* pregnant woman
* use of painkillers in the last twenty four hours
* presence of metal inside the head
* pacemaker
* wound on the area of electrodes' application
* drugs consumer
* recent application of transcranial direct stimulation
* psychiatric disease who lead the subject to a misunderstand of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold | Change in Pressure pain threshold just before the start of the intervention, immediately at the end of the intervention and 15 minutes after the end of the intervention
  Pressure pain threshold has been defined as the minimal amount of pressure at which a sense of pressure first changes to pain or discomfort

SECONDARY OUTCOMES:
Ability to generate motor images | Just before the start of the intervention
  The ability to generate motor images will be measured through The movement imagery questionnaire-revised (MIQ-R) is an 8-item self-report inventory that was used to assess visual and kinesthetic motor imagery ability. Four different movements are included in the MIQ-R, which is comprised of 4 visual and 4 kinesthetic items. For each item, participants read a description of the movement. They then physically performed the movement and were instructed to reassume the starting position after finishing the movement and before performing the mental task, imagining the movement visually or kinesthetically. Each participant then rated the ease or difficulty of mentally generating that image on a 7-point scale, in which 7 indicates "very easy to see/feel" and 1 "very difficult to see/feel." The internal consistencies of the MIQ-R have been consistently adequate.
Mental Chronometry | Just before the start of the intervention
  Mental chronometry is a reliable measure that has been widely used to record objective measurements of the ability to create mental motor images
The degree of physical activity | Just before the start of the intervention
  The level of physical activity will be assessed using the International Physical Activity Questionnaire, which allows the participants to be divided into 3 groups according to their level of activity, which can be high, moderate, and low or inactive

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No